CLINICAL TRIAL: NCT01062633
Title: Effect of Erythritol and Xylitol on Dental Caries Prevention in Children
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tartu (Other)
Collaborators: University of Turku (Other)
Responsible Party: Mare Saag prof, University of Tartu
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N012/95; VARST 07264 2008-2011
Record Dates: First submitted 2008-01-29; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2007-12

CONDITIONS: Dental Caries
Keywords: dental caries; prevention; dietary supplements
MeSH Terms: conditions — Dental Caries | interventions — Erythritol; Xylitol; Sorbitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A, observation (Experimental): dietary supplement
  Interventions: Dietary Supplement: A, erythritol
- B (Experimental): dietary supplement
  Interventions: Dietary Supplement: xylitol
- C (Experimental): dietary supplement
  Interventions: Dietary Supplement: C, sorbitol

INTERVENTIONS:
Dietary Supplement: A, erythritol — 2,5 g 3 times a day
  Arms: A, observation
Dietary Supplement: xylitol — 2,5 g 3 times a day
  Arms: B
Dietary Supplement: C, sorbitol — 2,5 g 3 times aday
  Arms: C

SUMMARY:
This study aims at demonstrating the effect of erythritol and xylitol lozenges on preventing the new caries lesions and the possible remineralization effect of both polyols on incipient caries lesions.

DETAILED DESCRIPTION:
Rationale: Several polyols (xylitol, sorbitol, erythritol) have been shown to act as excellent sugar substitutes, especially for in-between meals food products. Most commonly they are used in chewing gums, but the recent field trials also show a clear effectiveness of xylitol lozenges. Although sorbitol is metabolized at a slower rate than sucrose and not at all by most microorganisms, it can be fermented at a slow rate by all of the mutans streptococci including S. mutans while xylitol and erythritol are considered to be non-acidogenic. It has been demonstrated in some studies that xylitol reduces to a greater extent caries rate than sorbitol, however, the scientific committee on medicinal products is of the opinion that no clear data support the concept that xylitol possesses specific effects in vivo which validate a superiority claim over other polyols.

Objective: It is believed that the benefits of sugar-free gums may be twofold; 1) decreased lactic acid production and increased salivary flow potentially leading to an increased buffering of acids in plaque and 2) increased supersaturation of saliva with the mineral ions as well as enhanced clearance of sugars from the mouth. Thus sugar substitution and salivary stimulation could, it has been argued, be equally responsible for the noncariogenicity of sugar-free chewing gum. By comparing long term effects of several polyols, on possible remineralization effect on incipient caries lesions and on preventing the new caries lesions in comparison with sorbitol,the study will help demonstrate the superiority of erythritol and eventually xylitol over sorbitol and will help demonstrate the role of sugar substitutes, beyond saliva stimulation-mediated oral benefits on dental caries prevention.Sorbitol lozenges are used as a positive control. The saliva and plaque sample analyses would reveal the possible mechanisms of the expected caries preventive effects.

Study design: This is a double-blind, parallel, randomized, controlled study in primary school children around Tartu city. The allocation of the children into three groups will be based on classrooms for the practical reasons. The classrooms will be randomly allocated into the intervention and control groups. The study will last three years. During the first 2 years, the two intervention groups will consume either xylitol or erythritol-containing lozenges and the control group will be provided with sorbitol-containing tablets Then, there will be two options, depending on the effects on caries prevention after 2 years feeding with the polyols and depending on the SD of the caries incidence,. If the SD >2, the groups will not be spilt up as the power of the study would not be high enough to see any statistical effect. In this case, during the third experimental year, groups will stop eating polyol-containing lozenges and tablets to assess the lasting preventive effects of the polyol. If the SD<2 , the groups will be spilt up into two sub-groups, where one sub-group will stop eating polyols-containing lozenges to assess the lasting effect of polyol on caries prevention and the other sub-group will continue consuming the polyol-containing lozenges to assess the long-term effect of polyol intake on caries prevention.

Study population: The classrooms of 1st and 2nd primary schoolchildren (n=450) will be randomly allocated into two intervention groups (erythritol and xylitol) and into one positive control group (sorbitol. The list of the 1st and 2nd graders classrooms will be used as a sample frame. The allocation of the classrooms will be based on the random numbers generated by a computer.

Intervention: The test products will be distributed to the pupils in all (erythritol, xylitol, and sorbitol) groups three times a day during the school days (about 200/year) by the teachers.

Main study parameters/endpoints: All children will be clinically examined at the beginning of the trial, one -, two - and three years after the baseline examinations. All the surfaces of the mixed dentition (primary and permanent teeth) will be examined. The mean annual incipient and dentinal caries increment will be calculated. The teeth (FT) and surfaces (FS) restored or extracted because of caries during the study period will be calculated and included in the caries experience indices (dmft/DMFT). The plaque and saliva samples will be collected in each examination.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There will be clinical examinations and plaque sample collection of the study subjects four times in this study. Each examination will take about 15 min. No risks for the pupils can be expected from these examinations. The children will be given a toothbrush and toothpaste every 6 months. After the study examinations, pupils will be driven to a museum by bus.

ELIGIBILITY:
Inclusion Criteria:

* Children who's parents have signed and returned informed consent form

Exclusion Criteria:

* Any eating disorder
* Refuse to continue

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
caries reduction | 3 years

SECONDARY OUTCOMES:
Depression of oral microorganisms | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mare Saag, PhD, Principal Investigator — University of Tartu; Eino Honkala, PhD, Study Director — University of Turku, Institute of Dentistry; Kauko Mäkinen, PhD, Study Chair — University of Turku
Locations (1):
- Department of Stomatology, University of Tartu, Tartu, Estonia

REFERENCES:
- [Background] Makinen KK, Saag M, Isotupa KP, Olak J, Nommela R, Soderling E, Makinen PL. Similarity of the effects of erythritol and xylitol on some risk factors of dental caries. Caries Res. 2005 May-Jun;39(3):207-15. doi: 10.1159/000084800. PMID 15914983
- [Background] Isokangas P, Tiekso J, Alanen P, Makinen KK. Long-term effect of xylitol chewing gum on dental caries. Community Dent Oral Epidemiol. 1989 Aug;17(4):200-3. doi: 10.1111/j.1600-0528.1989.tb00611.x. PMID 2758793
- [Background] Makinen KK, Bennett CA, Hujoel PP, Isokangas PJ, Isotupa KP, Pape HR Jr, Makinen PL. Xylitol chewing gums and caries rates: a 40-month cohort study. J Dent Res. 1995 Dec;74(12):1904-13. doi: 10.1177/00220345950740121501. PMID 8600188
- [Background] Honkala E, Honkala S, Shyama M, Al-Mutawa SA. Field trial on caries prevention with xylitol candies among disabled school students. Caries Res. 2006;40(6):508-13. doi: 10.1159/000095650. PMID 17063022
- [Derived] Stsepetova J, Truu J, Runnel R, Nommela R, Saag M, Olak J, Nolvak H, Preem JK, Oopkaup K, Krjutskov K, Honkala E, Honkala S, Makinen K, Makinen PL, Vahlberg T, Vermeiren J, Bosscher D, de Cock P, Mandar R. Impact of polyols on Oral microbiome of Estonian schoolchildren. BMC Oral Health. 2019 Apr 18;19(1):60. doi: 10.1186/s12903-019-0747-z. PMID 30999906
- [Derived] Falony G, Honkala S, Runnel R, Olak J, Nommela R, Russak S, Saag M, Makinen PL, Makinen K, Vahlberg T, Honkala E. Long-Term Effect of Erythritol on Dental Caries Development during Childhood: A Posttreatment Survival Analysis. Caries Res. 2016;50(6):579-588. doi: 10.1159/000450762. Epub 2016 Nov 3. PMID 27806364
- [Derived] Honkala S, Runnel R, Saag M, Olak J, Nommela R, Russak S, Makinen PL, Vahlberg T, Falony G, Makinen K, Honkala E. Effect of erythritol and xylitol on dental caries prevention in children. Caries Res. 2014;48(5):482-90. doi: 10.1159/000358399. Epub 2014 May 21. PMID 24852946
- [Derived] Runnel R, Makinen KK, Honkala S, Olak J, Makinen PL, Nommela R, Vahlberg T, Honkala E, Saag M. Effect of three-year consumption of erythritol, xylitol and sorbitol candies on various plaque and salivary caries-related variables. J Dent. 2013 Dec;41(12):1236-44. doi: 10.1016/j.jdent.2013.09.007. Epub 2013 Oct 3. PMID 24095985
- [Derived] Runnel R, Honkala S, Honkala E, Olak J, Nommela R, Vahlberg T, Makinen KK, Saag M. Caries experience in the permanent dentition among first- and second-grade schoolchildren in southeastern Estonia. Acta Odontol Scand. 2013 May-Jul;71(3-4):410-5. doi: 10.3109/00016357.2012.690529. Epub 2012 May 21. PMID 22607272